CLINICAL TRIAL: NCT06809335
Title: A Pilot of a Personalized Circadian MHealth to Improve Sleep in Night Shift Workers
Acronym: SAIL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Philip Cheng, Associate Scientist, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16061
Record Dates: First submitted 2025-01-23; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Shift Work Sleep Disorder
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SHIFT App (Experimental): Participants in this condition will receive an access code to download the mobile application and conduct an orientation to SHIFT and the study procedures with a study team member. They will then enter four weeks of study directed use of SHIFT where they are trained on a daily procedure of opening SHIFT at the beginning of their day and planning their day in accordance with the app recommendations. App usage (4 times per week) will be incentivized with weekly bonuses added to study compensation. Following the four weeks of study-directed use, participants will continue with self-directed use. At four months, participants will then complete a booster session with two additional weeks of study-directed use, followed by self-directed use until the end of the study. The structure with the booster session has evidence for maintaining treatment gains and is also in alignment with the commercialization plan.
  Interventions: Other: Personalized circadian mHealth
- Waitlist Control (No Intervention): Participants in this condition will only complete questionnaires for the initial eight months. Those who remain shift workers will have the option of receiving the SHIFT app and the option to complete follow-up surveys in the same manner as the SHIFT App condition.

INTERVENTIONS:
Other: Personalized circadian mHealth — SHIFT is a mobile application designed to improve sleep in night shift workers. The SHIFT mobile application is used to collect data from an Apple Watch to assess an individual shift worker's body-clock timing and make personalized recommendations of light exposure schedules that are designed to align the body-clock with the night shift work schedule.
  Other Names: SHIFT
  Arms: SHIFT App

SUMMARY:
The goal of this project is to establish the evidence base for equitable accessibility and implementation of the precision sleep medicine mobile application, SHIFT.

ELIGIBILITY:
Inclusion Criteria:

* Inadequate sleep duration (habitual sleep less than 7 hours during the day)
* Willingness to download the SHIFT app and follow the lighting recommendations
* Ability to follow a set sleep schedule of 7 hours in bed after the night shifts
* Working at least 4 night shifts a month
* Shifts that must begin between 18:00 and 02:00 and last 8 to 12 hours
* Score of 8 or above on the Epworth Sleepiness scale and/or a score of 8 or above on the Insomnia Severity Index

Exclusion Criteria:

* Other independent sleep disorders (e.g., obstructive sleep apnea, narcolepsy, etc.)
* History of seizures or other significant neurological disorders
* Bipolar disorder
* Termination of shift schedule
* Pregnancy
* Current use of medications that impact sleep-wake functioning
* Alcohol and substance use disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Establish the effect of SHIFT on stakeholder-centered outcomes. | From enrollment to the 8 month point.
  Aim 1a. Measure the effect of SHIFT on work productivity and satisfaction compared to waitlist control using the Job Satisfaction Index. Effect will be tested using a mixed-effects linear regression model with participants as the random effect and Time, Condition, and the Time × Condition interaction term as the fixed effects.
  Aim 1b: Measure the effect of SHIFT on global health compared to waitlist control using the NIH PROMIS Global Health questionnaire. Effect will be tested using the same method as Aim 1a.
  Aim 1c. Measure the effect of SHIFT on turnover compared to waitlist control, measured at 8-month follow-up. Turnover will be operationalized as an individual who has either terminated the position they were in at baseline or is no longer engaged in shift work as operationalized in the study. Effect will be determined using a generalized mixed-effects regression with turnover as a dichotomous outcome.
Compare use experience and accuracy of SLEEP Android to the original iOS version. | From enrollment to the 8 month point.
  Aim 2a. Measure user experience of Android and iOS versions of SHIFT using the User Experience Questionnaire (UEQ). The following ranges of clinical indifference will be used: ± 3 points on the User Experience Questionnaire based on the bin size of 6 for each of the thresholds (bad, neutral, and good user experience).
  Aim 2b. Measure accuracy of predicted circadian misalignment (CM), sleep, and depression in Android and iOS versions. CM will be indexed with the outputs of the biomathematical model of the circadian system. Sleep will be measured using the Insomnia Severity Index and sleep diaries. Depression will be measured using the Quick Inventory of Depressive Symptomatology. The following ranges of clinical indifference will be used: 1) predicted CM = ± 3 hours based on approximately 2x the absolute mean error of our model predictions, 2) insomnia severity = ± 6 points, and 3) depression = 28.5% of the QIDS-SR16 score.

SECONDARY OUTCOMES:
Assess facilitators and barriers to engagement and implementation. | Immediately following completion of 8-month treatment period.
  A series of semi-structured interviews will be used for thematic analysis, and a comprehensive roadmap for future app updates based on user feedback. The semi-structured interviews will utilize the interview-guide approach following the CFIR framework selected for this study. Six phases will be followed for thematic analysis: (1) data familiarization, (2) generating initial codes, (3) searching for themes, (4) reviewing themes, (5) defining and naming themes, and (6) producing the report. We will combine deductive and inductive techniques to increase the accuracy of thematic analyses.

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Columbus Medical Center, Novi, Michigan, United States

IPD SHARING:
Plan to Share IPD: No